CLINICAL TRIAL: NCT06977958
Title: Efficacy of a 12-Week NASM Optimum Performance Training Program on Gluteal Muscle Strength, Hip Aesthetics, and Low Back Pain in Non-Athletic Women: A Randomized Controlled Trial
Brief Title: NASM OPT for Gluteal Enhancement in Non-Athletic Women: An RCT
Acronym: GlutealEnhan
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sistan and Baluchestan (Other)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, Assoc.Prof.Dr. of Sports Sciences, University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9378-30-2-2025
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain; Muscle Weakness; Body Image Disturbance
Keywords: NASM OPT; Gluteal Muscles; Hip Aesthetics; Non-Athletic Women; Resistance Training
MeSH Terms: conditions — Low Back Pain; Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blind (outcome assessors only; participants/instructors unblinded due to intervention nature).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NASM OPT Group (Experimental): Behavioral: NASM OPT Program Three 60-minute weekly sessions for 12 weeks, progressing through stabilization (weeks 1-4), strength endurance (weeks 5-8), and hypertrophy (weeks 9-12) phases. Exercises included hip thrusts, squats, and glute bridges.
  Interventions: Behavioral: NASM OPT Group
- General Exercise Group (Active Comparator): Behavioral: General Exercise Three 60-minute weekly sessions of brisk walking and light aerobics without targeted resistance training.
  Interventions: Behavioral: General Exercise Group

INTERVENTIONS:
Behavioral: NASM OPT Group — Three 60-minute weekly sessions for 12 weeks, progressing through stabilization (weeks 1-4), strength endurance (weeks 5-8), and hypertrophy (weeks 9-12) phases. Exercises included hip thrusts, squats, and glute bridges.
  Arms: NASM OPT Group
Behavioral: General Exercise Group — Three 60-minute weekly sessions of brisk walking and light aerobics without targeted resistance training.
  Arms: General Exercise Group

SUMMARY:
This RCT evaluates a 12-week NASM OPT program targeting gluteal muscle strength, hip aesthetics (shape, lift, circumference), and low back pain in 120 non-athletic women. The intervention group performed structured resistance training, while the control group engaged in general exercise. Outcomes included gluteal strength (dynamometer), aesthetic satisfaction (Likert scale), and functional performance (squat test).

DETAILED DESCRIPTION:
Participants were randomized to NASM OPT (3 weekly sessions: stabilization, strength, and hypertrophy phases) or general exercise (brisk walking/aerobics). Measurements at baseline and 12 weeks included gluteal strength, hip circumference, low back pain (VAS), and perceived aesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Non-athletic women (no exercise in prior 6 months).
* Interest in improving hip aesthetics.
* No musculoskeletal injuries.

Exclusion Criteria:

* Pregnancy
* Chronic illness
* Exercise contraindications

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Gluteal Strength | Baseline, 12 weeks (post-intervention)
  kg; handheld dynamometer
Perceived Hip Shape/Lift | Baseline, 12 weeks (post-intervention)
  5-point Likert scale
Hip Circumference | Baseline, 12 weeks (post-intervention)
  cm

SECONDARY OUTCOMES:
Aesthetic Satisfaction | Baseline, 12 weeks
  5-point Likert scale
Functional Performance | Baseline, 12 weeks
  30-second squat test
Low Back Pain | Baseline, 12 weeks
  VAS, 0-10 cm

CONTACTS AND LOCATIONS:
Overall Officials: Mohammadreza Rezaeipour, MD, PhD, Study Director — Assoc.Prof.Dr. of University of Sistan and Baluchestan, Zahedan, Iran
Locations (1):
- Ferdows Shafa Center, Ferdows, South Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: No
Privacy concerns regarding sensitive participant data.